CLINICAL TRIAL: NCT01717456
Title: Conservative Treatment of Fecal Incontinence: Community-Based Effectiveness Trial
Brief Title: Educational-Medical-Behavioral Treatment of Fecal Incontinence
Acronym: FIX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment led sponsor to terminate study early.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, William (Bill) Whitehead, PhD, Professor of Medicine and Adjunct Professor of OBGYN, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-1569; R01HS018695 (AHRQ)
Record Dates: First submitted 2012-09-15; First posted 2012-10-30 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Fecal Incontinence
Keywords: Fecal incontinence; Frail elders; Home health care; Nurse; Patient education
MeSH Terms: conditions — Fecal Incontinence | interventions — Educational Status; Laxatives; Loperamide; polyethylene glycol 3350; Polyethylene Glycols; Clothing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational-Medical-Behavioral (Active Comparator): Educational-Medical-Behavioral intervention includes education, fiber supplements [Metamucil 1-4 packets (3.4-13.6 g)/day], laxatives or anti-diarrheals [Miralax 1-2 packets (17-34 g)/day or Imodium 0.5-2 tablets (1-4 mg)/day], pelvic floor muscle exercises [100 10-second squeezes/day], tips on how to prevent fecal incontinence, daily diary, and protective pads or garments [as needed].
  Interventions: Other: Education; Dietary Supplement: Fiber supplements; Drug: Laxatives or anti-diarrheals; Behavioral: Pelvic floor muscle exercises; Behavioral: Tips on how to prevent fecal incontinence; Behavioral: Daily diary; Other: Protective pads or garments
- Standard Care (Placebo Comparator): Standard care includes fiber supplements 1-4 packets (3.4-13.6 g)/day], daily diary, and protective pads or garments [as needed].
  Interventions: Dietary Supplement: Fiber supplements; Behavioral: Daily diary; Other: Protective pads or garments

INTERVENTIONS:
Other: Education — Patient and caregiver will be taught which muscles are used in continence and defecation through the use of a training manual and anatomical drawings.
  Arms: Educational-Medical-Behavioral
Dietary Supplement: Fiber supplements — Patients and caregivers will be taught to use fiber supplements to normalize stool consistency if patient reports diarrhea or constipation. Fiber supplements will be in the form of Metamucil beginning with 3.4 grams per day and increasing up to 13.6 grams per day if needed to control stool consistency.
Drug: Laxatives or anti-diarrheals — Miralax at a dose of one packet (17 grams) daily may be used for constipation if unresponsive to fiber. Dose may be titrated up to two packets (34 grams) daily if needed.
  Imodium at a starting dose of 2 mg/day may be used for diarrhea if unresponsive to fiber. Dose of Imodium may be titrated down to 1 mg or up to 4 mg if needed.
  Other Names: Miralax (polyethylene glycol); Imodium (loperamide)
  Arms: Educational-Medical-Behavioral
Behavioral: Pelvic floor muscle exercises — Patients will be taught how to perform pelvic floor muscle contractions during digital rectal examination by a nurse. They will be asked to squeeze 100 times daily.
  Arms: Educational-Medical-Behavioral
Behavioral: Tips on how to prevent fecal incontinence — Examples of behavioral tips are "Walk, don't run to the toilet" and "Squeeze before you lift objects or sneeze".
  Arms: Educational-Medical-Behavioral
Behavioral: Daily diary — Both groups will keep a daily diary, but amount of detail differs: Active comparator group records bowel accidents, bowel movements, Bristol Stool ratings of stool consistency, number of times they do pelvic floor exercises, study medications, and comments for the nurse to read. Placebo comparator group records only bowel accidents, bowel movements, and Bristol Stool scores.
Other: Protective pads or garments — In both groups, patients will be permitted to use pads or protective garments to avoid embarrassment. They will be told that fecal leakage that is stopped by a pad or protective garment should still be recorded as fecal incontinence.
  Other Names: Continence pads

SUMMARY:
In previous studies at a university referral center the investigators demonstrated that a multicomponent conservative treatment for fecal incontinence was effective. The treatment combines patient education with medical management of diarrhea and constipation plus behavioral training. The purpose of this study is to determine whether this treatment is effective when delivered by home health care nurses to frail elderly patients.

DETAILED DESCRIPTION:
Fecal incontinence (FI) affects 9% of U.S. adults and occurs weekly or more often in 2.7%. Prevalence increases with age reaching 15% by 70 years. FI has a devastating impact on quality of life and substantially increases caregiver burden when patients have comorbid conditions requiring caregiver assistance. The investigators propose an effectiveness trial whose overall goal is to determine whether a conservative intervention which has been shown to be effective in single-site studies will sustain its efficacy when disseminated to a home bound population by home health care nurses. The treatment includes patient education about the physiology of how continence is maintained, pelvic floor exercises, behavioral strategies for preventing FI, and use of fiber or nonprescription medication to treat diarrhea or constipation. To minimize drift when the treatment is disseminated to a large group of providers, patient education and other basic components of treatment are included in a printed training manual and are available to nurse providers on a website; however, nurse supervision to individualize treatment remains important. The study will be carried out in 8 counties in central North Carolina which are served by the University of North Carolina Home Health Care and Rex Home Health Care agencies (partners in this study). Nurses in these agencies will be randomly assigned to two groups. For the first two years all patients of the nurses in one group will receive the active intervention while all patients of nurses in the other group will receive usual care plus a training manual and symptom monitoring to control for expectancy. After two years, all patients in these home health care agencies will receive the active intervention. After excluding patients with severe cognitive impairment and those with stomas, the investigators estimate 252 - 340 patients with FI who are over age 50 will receive treatment (at least 189 in active treatment and 63 controls). Specific aims are (1) to show that the active treatment is more effective than the control treatment for improving FI severity, patient quality of life, and caregiver burden, and that improvements are maintained for at least 6 months; (2) to identify moderators of treatment effectiveness (candidate variables are cognitive status, mobility impairment, willingness of family caregiver to assist with treatment, anxiety, depression, age, and race); and (3) to explore whether successful treatment of FI reduces the risk of nursing home referral.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported fecal incontinence at least once a month
* Family caregiver available and willing to participate in treatment sessions and willing to assist patient with study procedures
* Patients and caregivers willing to be interviewed by a research assistant in their home on three occasions
* Onset of fecal incontinence more than 3 months previously (i.e., not transient fecal incontinence)

Exclusion Criteria:

* Has a stoma or fecal incontinence status is unknown
* Has fecal incontinence less than monthly
* Severe cognitive impairment (response of 4 on OASIS question M1700)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William E Whitehead, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Insufficient data to be analyzed by an outside investigator.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Home Health Care (HHC) provided lists to the investigators of new patients who were screened by HHC using the OASIS Questionnaire. Research assistants identified eligible patients based on the OASIS questions and telephoned them to obtain verbal consent and to schedule a baseline assessment visit. Written consent was obtained at the baseline visit.
Pre-assignment Details: Baseline data collection and written consent was obtained at a home visit prior to referring the patient to HHC for randomization and initiation of treatment. Only 19/31 who gave consent to the research assistant were randomized. 3 others were judged ineligible by HHC, and 9 dropped out while awaiting treatment.
Period: End of Treatment
Arm/Group | Educational-Medical-Behavioral | Standard Care
Started | 11 | 8
Completed | 11 | 6
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Follow-Up 6 Months After End of Tx
Arm/Group | Educational-Medical-Behavioral | Standard Care
Started | 11 | 6
Completed | 7 | 2
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is limited to patients who were randomized after referral to Home Health Care.
Groups:
- Educational-Medical-Behavioral: Educational-Medical-Behavioral intervention includes education, fiber supplements [Metamucil 1-4 packets (3.4-13.6 g)/day], laxatives [mirilax 1-2 packets or 17-34 g/day] or anti-diarrheal medication [Imodium 1-4 mg/day], pelvic floor muscle exercises [100 10-second squeezes/day], tips on how to prevent fecal incontinence, and use of a daily diary and protective pads or garments [if needed].
- Total: Total of all reporting groups
Arm/Group | Educational-Medical-Behavioral | Standard Care | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 86.11 (4.51) | 85.00 (3.61) | 85.83 (4.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 3 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 5 | 5
Fecal Incontinence Severity Index (FISI) at Baseline [Mean (Standard Deviation); unit: units on a scale] — Subjects rated the frequency of 4 types of stool leakage (gas, mucus, liquid, and solid) over the prior month on a 6-stepscale. Possible responses were never, 1-3 times/ month, once/week, 2 or more times/week, once/day, and 2 or more times/day. Based on the average quality of life impact scores assigned by a reference group of 34 subjects with fecal incontinence, weights were assigned to each of these 4 responses and added together for a sum score. Range is 0-61. No guidance on what defines mild, moderate, or severe is available. Higher scores show more severe fecal incontinence.
  units on a scale | 24.50 (12.22) | 22.75 (8.14) | 23.72 (2.44)
Manchester Health Questionnaire (MHQ) Severity Scale at Baseline [Mean (Standard Deviation); unit: units on a scale] — The MHQ (Br J Obstetrics & Gynecol 2001;108:1057-67) is a 32-item questionnaire that assesses the impact of anal incontinence on quality of life in women. Each item is answered on a 5-point ordinal scale. Eight of 9 subscales were used: incontinence impact, role, physical function, social function, personal function, emotional problems, sleep/energy, and severity. A total score was calculated by summing the subscales. The range of scores of each domain is 0-100, and higher scores indicate greater impairment. Means and SDs for a reference group of 154 FI patients were published.
  units on a scale | 48.64 (17.76) | 50.00 (18.13) | 49.21 (17.42)
MHQ Incontinence Impact at Baseline [Mean (Standard Deviation); unit: units on a scale] — The MHQ (Br J Obstetrics & Gynecol 2001;108:1057-67) is a 32-item questionnaire that assesses the impact of anal incontinence on quality of life in women. Each item is answered on a 5-point ordinal scale. Eight of 9 subscales were used: incontinence impact, role, physical function, social function, personal function, emotional problems, sleep/energy, and severity. A total score was calculated by summing the subscales. This subscale has a range of 0-100, with higher scores signifying greater impairment in quality of life.
  units on a scale | 52.27 (23.60) | 65.63 (26.52) | 57.89 (25.07)
MHQ Role Limitations at Baseline [Mean (Standard Deviation); unit: units on a scale] — The MHQ (Br J Obstetrics & Gynecol 2001;108:1057-67) is a 32-item questionnaire that assesses the impact of anal incontinence on quality of life in women. Each item is answered on a 5-point ordinal scale. Eight of 9 subscales were used: incontinence impact, role, physical function, social function, personal function, emotional problems, sleep/energy, and severity. A total score was calculated by summing the subscales. This subscale has a range of 0-100, with higher scores signifying greater impairment in quality of life.
  units on a scale | 13.64 (26.49) | 50.00 (29.12) | 28.95 (32.56)
MHQ Physical Limitations at Baseline [Mean (Standard Deviation); unit: units on a scale] — The MHQ (Br J Obstetrics & Gynecol 2001;108:1057-67) is a 32-item questionnaire that assesses the impact of anal incontinence on quality of life in women. Each item is answered on a 5-point ordinal scale. Eight of 9 subscales were used: incontinence impact, role, physical function, social function, personal function, emotional problems, sleep/energy, and severity. A total score was calculated by summing the subscales. This subscale has a range of 0-100, with higher scores signifying greater impairment in quality of life.
  units on a scale | 18.18 (21.91) | 50.00 (28.35) | 31.58 (28.98)
MHQ Social Limitations at Baseline [Mean (Standard Deviation); unit: units on a scale] — The MHQ (Br J Obstetrics & Gynecol 2001;108:1057-67) is a 32-item questionnaire that assesses the impact of anal incontinence on quality of life in women. Each item is answered on a 5-point ordinal scale. Eight of 9 subscales were used: incontinence impact, role, physical function, social function, personal function, emotional problems, sleep/energy, and severity. A total score was calculated by summing the subscales. This subscale has a range of 0-100, with higher scores signifying greater impairment in quality of life.
  units on a scale | 16.67 (29.11) | 43.75 (35.57) | 28.07 (33.93)
MHQ Personal Relationships at Baseline [Mean (Standard Deviation); unit: units on a scale] — The MHQ (Br J Obstetrics & Gynecol 2001;108:1057-67) is a 32-item questionnaire that assesses the impact of anal incontinence on quality of life in women. Each item is answered on a 5-point ordinal scale. Eight of 9 subscales were used: incontinence impact, role, physical function, social function, personal function, emotional problems, sleep/energy, and severity. A total score was calculated by summing the subscales. This subscale has a range of 0-100, with higher scores signifying greater impairment in quality of life.
  units on a scale | 8.33 (20.41) | 20.00 (32.60) | 13.64 (25.89)
MHQ Emotions at Baseline [Mean (Standard Deviation); unit: units on a scale] — The MHQ (Br J Obstetrics & Gynecol 2001;108:1057-67) is a 32-item questionnaire that assesses the impact of anal incontinence on quality of life in women. Each item is answered on a 5-point ordinal scale. Eight of 9 subscales were used: incontinence impact, role, physical function, social function, personal function, emotional problems, sleep/energy, and severity. A total score was calculated by summing the subscales. This subscale has a range of 0-100, with higher scores signifying greater impairment in quality of life.
  units on a scale | 19.70 (15.49) | 51.04 (28.67) | 32.89 (26.57)
MHQ Sleep Energy at Baseline [Mean (Standard Deviation); unit: units on a scale] — The MHQ (Br J Obstetrics & Gynecol 2001;108:1057-67) is a 32-item questionnaire that assesses the impact of anal incontinence on quality of life in women. Each item is answered on a 5-point ordinal scale. Eight of 9 subscales were used: incontinence impact, role, physical function, social function, personal function, emotional problems, sleep/energy, and severity. A total score was calculated by summing the subscales. This subscale has a range of 0-100, with higher scores signifying greater impairment in quality of life.
  units on a scale | 7.95 (14.00) | 23.44 (28.69) | 14.47 (22.15)
Zarit Caregiver Burden Scale at Baseline [Mean (Standard Deviation); unit: units on a scale] — The Zarit Caregiver Burden Interview is a 22-item questionnaire to assess the perceived burden of taking care of another ill or physically impaired person. All items are answered on a 5-step ordinal scale (from never to nearly always). Higher scores depict greater burden on the family. The total score range is from 0 to 66.
  units on a scale | 36.00 (42.43) | 18.33 (13.50) | 22.75 (14.13)
Frequency of fecal incontinence at Baseline [Median (Full Range); unit: units on a scale] — OASIS question M1620. 6-level ordinal scale.
  0 = Never or rarely incontinent for stool
  1. = Less than 1/week
  2. = 1-3 days/week
  3. = 4-6 days/week
  4. = Daily stool leakage
  5. = Multiple times per day
  Higher scores represent worse outcomes.
  Data were missing for 2/11 in Group A and for 6/8 in Group B. Population: Data were missing for 2/11 in Group A and 6/8 in Group B.
  units on a scale
    number analyzed (Participants) | 9 | 2 | 11
    (all) | 2 [1 to 5] | 4.5 [4 to 5] | 2 [1 to 5]
Urinary Continence Status at Baseline [Median (Full Range); unit: units on a scale] — OASIS Question M1610 is a 3-level ordinal scale.
  0 = No urinary incontinence
  1. = Incontinence for urine
  2. = Patient requires catheter
  Data are missing for 2/11 in Group A and 6/8 in Group B. Having a catheter is equivalent to having urinary incontinence; therefore, the investigators treated a 2 as equivalent to a 1. Population: Data were missing for 2/11 in Group A and 6/8 for Group B.
  units on a scale
    number analyzed (Participants) | 9 | 2 | 11
    (all) | 1 [0 to 1] | 0.5 [0 to 1] | 1 [0 to 1]
Cognitive Function at Baseline [Median (Full Range); unit: units on a scale] — OASIS Question M1700. 5-level ordinal scale:
  0 = Alert and oriented
  1. = Requires prompting for unfamiliar activities
  2. = Requires assistance when task demands shifting attention
  3. = Requires assistance for routine tasks
  4. = Totally dependent
  Data missing for 2/11 in Group A and 6/8 in Group B. A higher number indicates a greater degree of cognitive impairment. Population: Data were missing for 2/11 in Group A and 6/8 for Group B.
  units on a scale
    number analyzed (Participants) | 9 | 2 | 11
    (all) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Ambulation at Baseline [Median (Full Range); unit: units on a scale] — OASIS Question M1860 is a 7-level ordinal scale.
  0 = Walks without assistance
  1. = Uses cane or other one-hand assistive device
  2. = Uses walker or other two-hand assistive device
  3. = Able to walk with assistance
  4. = Chair-fast but can wheel self around
  5. = Chair-fast and requires assistance
  6. = Bedfast
  Higher scores indicate a greater degree of physical impairment.
  units on a scale | 0 [0 to 2] | 0.5 [0 to 1] | 0.2 [0 to 2]
Ability to use toilet at Baseline [Median (Full Range); unit: participants] — OASIS Question M1840 is a 5 level ordinal scale. Steps are:
  0 = Independent self-toileting
  1. = Uses toilet when reminded to do so
  2. = Unable to reach toilet but can use a bedside commode
  3. = Limited to use of a bedpan
  4. = Totally dependent in toileting
  Missing data for 2/11 in Group A and 6/8 in Group B.
  Higher scores indicate a greater degree of impairment in toileting behavior. Population: Data were missing for 2/11 in Group A and 6/8 for Group B.
  participants
    number analyzed (Participants) | 9 | 2 | 11
    (all) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
When is patient anxious at Baseline? [Median (Full Range); unit: units on a scale] — OASIS Question M1720 is a 4-level ordinal scale. Responses are:
  0 = Never
  1. = Less than every day
  2. = Daily but not constantly
  3. = All the time
  Higher scores indicate a greater level of anxiousness.
  units on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Depression Screening at Baseline [Number; unit: participants] — OASIS Question M1730 has 4 discrete categories. Possible responses are:
  0 = Patient was not screened for depression
  1. = Screened by PHQ2 depression scale
  2. = Meets criteria for further screening for depression
  3. = Does not meet criteria for further screening
  Higher scores indicate a greater level of depression.
  participants
    Not screened for depression | 8 | 1 | 9
    Screened by Patient Health Questionnaire 2 (PHQ2) | 1 | 1 | 2
    Requires further evaluation | 0 | 0 | 0
    Screened and does not need further evaluation | 0 | 0 | 0
    Unknown | 2 | 6 | 8
Living Situation at Baseline [Number; unit: participants] — OASIS Question M1100 has 3 discrete categories which are:
  1 = Lives alone 6 = Lives with another person 11 = Lives in assisted living
  Scores are labels describing the patient's living situation.
  participants
    Lives alone | 3 | 0 | 3
    Lives with another adult | 4 | 2 | 6
    Lives in assisted living | 2 | 0 | 2
    Unknown | 2 | 6 | 8
Source of Assistance with ADLs at Baseline [Number; unit: participants] — OASIS Question M2100 has 5 discrete categories which are:
  0 = No assistance needed
  1. = Caregiver provides assistance for activities of daily living (ADLs)
  2. = Caregiver needs training or support
  3. = Caregiver is not likely to provide assistance
  4. = Unclear if caregiver will provide assistance
  5. = Assistance needed but none is available
  Higher scores indicate a greater need for assistance with ADLs.
  participants
    No assistance needed | 5 | 2 | 7
    Caregiver provides assistance | 3 | 0 | 3
    Caregiver needs training or support | 0 | 0 | 0
    Caregiver unlikely to provide assistance | 0 | 0 | 0
    Unclear if caregiver will assist patient | 0 | 0 | 0
    Assistance needed but not available | 0 | 0 | 0
    Unknown | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Fecal Incontinence Severity Index (FISI) at End of Treatment
Description: At the end of treatment, the FISI requires the patient to report the frequency of occurrence of 4 types of fecal incontinence (solid, liquid, mucus, and gas incontinence) in the past month. These four responses are multiplied by empirically derived patient weights and the values are added together. Range of scores is 0-61. Higher scores show more severe fecal incontinence.
Time Frame: End of Treatment (Week 6)
Population: Analysis population includes all participants who provided end of treatment data to research assistants during a home visit. One subject from the EMB treatment did not provide data, and 1 subject from the SC group did not provide these data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 10 | 5
units on a scale | 18.00 (10.30) | 22.00 (9.17)
Statistical Analysis 1: Comparison: Educational-Medical-Behavioral vs Standard Care; Test type: Superiority or Other; p = .05, t-test, 2 sided — No adjustment for multiple comparisons; Mean Difference (Final Values) = 4.0, Standard Deviation 6.72

2. Primary Outcome: Fecal Incontinence Severity Index (FISI) at Follow-Up (FU)
Description: At follow up 6 months after the end of treatment, the subject reports the frequency of occurrence of 4 types of fecal incontinence (solid, liquid, mucus, and gas incontinence) in the past month. These four responses are multiplied by empirically derived patient weights and the values are added together. Range is 0-61. No data is available to interpret the scale as mild, moderate, or severe fecal incontinence.
Time Frame: 6 months after (6-Week) treatment ends
Population: The analysis sample consists of all patients who provided data at the 6 month FU visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 7 | 2
units on a scale | 14.86 (12.71) | 37.00 (21.21)

3. Secondary Outcome: Adequate Relief of Fecal Incontinence at End of Treatment
Description: At the end of treatment, the subject is asked, "Compared to before you started home health care, have you experienced adequate relief of your fecal incontinence symptoms? [Responses: yes or no]". A responder is anyone answering yes. A treatment would be judged successful if there was at least 10% more responders in the active compared to the control groups.
Time Frame: End of Treatment (Week 6)
Population: Data not available for 1/11 Educational-Medical-Behavioral group subject and for 2/8 Standard Care subjects.
Measure: Number; unit: participants
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 10 | 6
participants
  Yes, Adequate Relief | 5 | 1
  No, No Adequate Relief | 5 | 3
  Unknown | 0 | 2

4. Secondary Outcome: Adequate Relief of Fecal Incontinence at Follow Up
Description: At follow up 6 months after the end of treatment, the subject is asked, "Compared to before you started home health care, have you experienced adequate relief of your fecal incontinence symptoms? [Responses: yes or no]". A responder to treatment is a subject who answers "yes". When applied to group analysis, a treatment is regarded as effective if the responder rate is at least 10% greater in the active treatment arm compared to the control arm. This measure is not recorded at baseline because it is undefined until treatment has been provided.
Time Frame: 6 months after (6-Week) treatment ends
Population: Data not available for 3/7 Educational-Medical-Behavioral group subject and for 2/2 Standard Care subjects.
Measure: Number; unit: participants
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 7 | 2
participants
  Yes, Adequate Relief | 1 | 0
  No, no Adequate Relief | 3 | 0
  Unknown | 3 | 2

5. Secondary Outcome: MHQ Severity Scale at End of Treatment
Description: Quality of life scale specific to fecal incontinence. Severity is one of 8 MHQ subscales. This subscale has a range of 0 to 100. Higher scores indicate greater severity of QOL impact.
Time Frame: End of Treatment (Week 6)
Population: All subjects completing end of treatment home visit with research assistant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 11 | 8
units on a scale | 42.50 (28.41) | 55.00 (23.72)

6. Secondary Outcome: MHQ Severity Scale at Follow Up
Description: Quality of life scale specific to fecal incontinence. This is one of 8 subscales. This subscale has a range of 0 to 100. Higher scores indicate greater impact on quality of life.
Time Frame: 6 months after (6-Week) treatment ends
Population: All subjects completing end of treatment home visit with research assistant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 7 | 2
units on a scale | 39.29 (25.40) | 47.50 (31.82)

7. Secondary Outcome: Zarit Caregiver Burden Scale at End of Treatment
Description: Validated questionnaire developed to assess the psychosocial and health burden experienced by a family caregiver of the identified patient. The 22-items ask about behaviors and feelings of caregivers on a 6-step ordinal scale (never to almost always). The scale is valid for caregivers of individuals with diverse chronic disabilities (dementia, advanced cancer, acquired brain injury). The scale has good internal consistency. Total scores range 0-66, and 21 or greater is interpreted as high burden (J Clin Epidemiol 2010;63:535-42). Subscales (role and personal strain) have been described but are unreliable so total scores were used.
Time Frame: End of Treatment (Week 6)
Population: Family caregivers of patients completing the study. Some caregivers declined or no caregiver was available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 2 | 2
units on a scale | 33.00 (42.43) | 30.50 (23.34)

8. Secondary Outcome: Zarit Caregiver Burden Scale at Follow Up
Description: Validated questionnaire developed to assess the psychosocial and health burden experienced by a family caregiver of the identified patient. The total score range is from 0 to 66. Higher scores indicate greater severity of burden on the family.
Time Frame: 6 months after (6-Week) treatment ends
Population: Family caregivers of patients completing the study. Some caregivers declined or no caregiver was available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 7 | 2
units on a scale | 14.00 (14.00) | 25.50 (20.51)

9. Secondary Outcome: Fecal Incontinence Frequency at End of Treatment
Description: OASIS question M1620: Bowel incontinence frequency. Response options are:
  0 - Very rarely or never has bowel incontinence
  1. - Less than once weekly
  2. - One to three times weekly
  3. - Four to six times weekly
  4. - On a daily basis
  5. - More often than once daily
Time Frame: End of Treatment (Week 6)
Population: Analysis population consists of all patients who provided data at the end of treatment visit. Data is missing for 2/11 in Group A and 6/8 in Group B.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 9 | 2
units on a scale | 1 [0 to 3] | 2 [0 to 4]

10. Secondary Outcome: Urinary Incontinence Status Change From Baseline to End of Treatment
Description: OASIS question M1610: Urinary incontinence or urinary catheter presence. Response options are:
  0 - No incontinence or catheter (includes anuria or ostomy for urinary drainage)
  1. - Patient is incontinent
  2. - Patient requires a urinary catheter (i.e., external, indwelling, intermittent, suprapubic)
Time Frame: Baseline, end of treatment (week 6)
Population: Analysis population consists of all patients who provided end of treatment data. Data were missing for 2/11 in Group A and 6/8 in Group B.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 9 | 2
units on a scale | 1 [0 to 1] | 0.50 [0 to 1]

11. Secondary Outcome: Admission to Nursing Home at End of Treatment
Description: Was patient admitted to a nursing home for one or more days at any time between enrollment and follow-up 7-8 months after treatment onset.
Time Frame: End of Treatment (Week 6)
Population: Analysis sample was all patients who provided data at end of treatment.
Measure: Number; unit: participants
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 8 | 2
participants
  Admitted to nursing home | 0 | 0
  Not admitted to nursing home | 8 | 2

12. Secondary Outcome: MHQ Incontinence Impact at End of Treatment
Description: Quality of life scale specific to fecal incontinence. This is one of 8 subscales. This subscale has a range of 0-100, with higher scores signifying greater impairment in quality of life.
Time Frame: End of Treatment (Week 6)
Population: All subjects completing end of treatment home visit with research assistant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 10 | 5
units on a scale | 42.50 (23.72) | 70.00 (20.92)

13. Secondary Outcome: MHQ Incontinence Impact at Follow Up
Description: as for outcome 12
Time Frame: 6 months after (6-Week) treatment ends
Population: All subjects completing end of treatment home visit with research assistant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 7 | 2
units on a scale | 35.71 (24.40) | 25.00 (0.00)

14. Secondary Outcome: MHQ Role Limitations at End of Treatment
Description: as for outcome 12
Time Frame: End of Treatment (Week 6)
Population: All subjects completing end of treatment home visit with research assistant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 11 | 8
units on a scale | 16.25 (28.90) | 57.50 (34.91)

15. Secondary Outcome: MHQ Role Limitations at Follow Up
Description: as for outcome 12
Time Frame: 6 months after (6-Week) treatment ends
Population: All subjects completing end of treatment home visit with research assistant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 7 | 2
units on a scale | 14.29 (19.67) | 12.50 (17.68)

16. Secondary Outcome: MHQ Physical Limitations at End of Treatment
Description: as for outcome 12
Time Frame: End of Treatment (Week 6)
Population: All subjects completing end of treatment home visit with research assistant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 11 | 8
units on a scale | 18.75 (31.87) | 60.00 (32.36)

17. Secondary Outcome: MHQ Physical Limitations at Follow Up
Description: as for outcome 12
Time Frame: 6 months after (6-Week) treatment ends
Population: All subjects completing end of treatment home visit with research assistant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 7 | 2
units on a scale | 7.14 (18.90) | 31.25 (8.84)

18. Secondary Outcome: MHQ Social Limitations at End of Treatment
Description: as for outcome 12
Time Frame: End of Treatment (Week 6)
Population: All subjects completing end of treatment home visit with research assistant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 11 | 8
units on a scale | 15.83 (26.77) | 48.33 (43.46)

19. Secondary Outcome: MHQ Social Limitations at Follow Up
Description: as for outcome 12
Time Frame: 6 months after (6-Week) treatment ends
Population: All subjects completing end of treatment home visit with research assistant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 7 | 2
units on a scale | 2.38 (6.30) | 4.17 (5.89)

20. Secondary Outcome: MHQ Personal Relationships at End of Treatment
Description: as for outcome 12
Time Frame: End of Treatment (Week 6)
Population: All subjects completing end of treatment home visit with research assistant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 11 | 6
units on a scale | 0 (0) | 25.00 (35.36)

21. Secondary Outcome: MHQ Personal Relationships at Follow Up
Description: as for outcome 12
Time Frame: 6 months after (6-Week) treatment ends
Population: All subjects completing end of treatment home visit with research assistant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 7 | 2
units on a scale | 0 (0) | 0 (0)

22. Secondary Outcome: MHQ Emotions at End of Treatment
Description: as for outcome 12
Time Frame: End of Treatment (Week 6)
Population: All subjects completing end of treatment home visit with research assistant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 11 | 8
units on a scale | 24.17 (29.52) | 50.00 (38.64)

23. Secondary Outcome: MHQ Emotions at Follow Up
Description: as for outcome 12
Time Frame: 6 months after (6-Week) treatment ends
Population: All subjects completing end of treatment home visit with research assistant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 7 | 2
units on a scale | 13.10 (13.49) | 12.50 (5.89)

24. Secondary Outcome: MHQ Sleep Energy at End of Treatment
Description: as for outcome 12
Time Frame: End of Treatment (Week 6)
Population: All subjects completing end of treatment home visit with research assistant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 11 | 8
units on a scale | 10.00 (17.48) | 32.50 (20.92)

25. Secondary Outcome: MHQ Sleep Energy at Follow Up
Description: as for outcome 12
Time Frame: 6 months after (6-Week) treatment ends
Population: All subjects completing end of treatment home visit with research assistant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 7 | 2
units on a scale | 3.57 (6.10) | 0 (0)

26. Other Pre Specified Outcome: Cognitive Status at End of Treatment
Description: OASIS question M1700: Cognitive functioning: Patient's current (day of assessment) level of alertness, orientation, comprehension, concentration, and immediate memory for simple commands. Measure as treatment moderator. Response categories are:
  0 - Alert/oriented, able to focus and shift attention, comprehends and recalls task directions independently.
  1. - Requires prompting (cuing, repetition, reminders) only under stressful or unfamiliar conditions.
  2. - Requires assistance and some direction in specific situations (e.g., on all tasks involving shifting of attention), or consistently requires low stimulus environment due to distractibility.
  3. - Requires considerable assistance in routine situations. Is not alert and oriented or is unable to shift attention and recall directions more than half the time.
  4. - Totally dependent due to disturbances uch as constant disorientation, coma, persistent vegetative stte, or delirium.
Time Frame: End of Treatment (Week 6)
Population: Analysis population is all patients who provided data on this measure at end of treatment. Data were missing for 2/11 in Group A and 6/8 in Group B.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 9 | 2
units on a scale | 0 [0 to 1] | 0 [0 to 0]

27. Other Pre Specified Outcome: Change in Ambulation From Baseline to End of Treatment
Description: OASIS question M1860: Ambulation/locomotion: Current ability to walk safely, once in a standing position, or use a wheelchair, once in a seated position, on a variety of surfaces. Measure as a moderator of treatment effects. Responses:
  0. Able to independently walk on even and uneven surfaces and negotiate stairs with or without railings (i.e., needs no human assistance or assistive device).
  1. Requires use of a device (e.g., cane, walker) to walk alone or requires human supervision or assistance to negotiate stairs or steps or uneven surfaces.
  2. Able to walk only with the supervision or assistance of another person at all times.
  3. Chairfast, unable to ambulate but is able to wheel self independently.
  4. Chairfast, unable to ambulate and is unable to wheel self.
  5. Bedfast, unable to ambulate or be up in a chair.
  Higher scores represent improvement in ability to ambulate.
Time Frame: Baseline, End of Treatment (Week 6)
Population: Analysis sample consists of all patients who provided data for this questionnaire at the end of treatment. Two EMB subjects did not provide this data for unknown reasons, and 4 SC subjects did not provide this data for unknown reasons.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 9 | 2
units on a scale | 0 [0 to 2] | 0 [0 to 0]

28. Other Pre Specified Outcome: Ability to Reach Toilet at End of Treatment
Description: OASIS question M1840: Toilet transferring: Current ability to get to and from the toilet or bedside commode safely and transfer on and off toilet/commode. Measure as moderator of treatment outcomes.
  A lower score is better.
  Responses:
  0. Able to get to and from the toilet and transfer independently with or without a device.
  1. When reminded, assisted, or supervised by another person, able to get to and from the toilet.
  2. Unable to get to and from the toilet but is able to use a bedside commode (with or without assistance).
  3. Unable to get to and from the toilet or bedside commode but is able to use a bedpan/urinal independently.
  4. Is totally dependent in toileting.
Time Frame: End of Treatment (Week 6)
Population: All patients who provided data for this measure at the end of treatment.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 9 | 2
units on a scale | 0 [0 to 0] | 0 [0 to 0]

29. Other Pre Specified Outcome: When is Patient Anxious at End of Treatment?
Description: OASIS question M1720: When anxious (reported or observed within the last 14 days). Measured as moderator of treatment effects on ordinal scale. Higher scores indicate a greater level of anxiousness. Responses are:
  0 - None of the time
  1. - Less often than daily
  2. - Daily, but not constantly
  3. - All of the time
Time Frame: End of Treatment (Week 6)
Population: Analysis population consists of all patients who provided end of treatment data.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 9 | 2
units on a scale | 0 [0 to 0] | 0 [0 to 0]

30. Other Pre Specified Outcome: Depression Screening at End of Treatment
Description: OASIS question M1730: Depression Screening. Measure as a moderator of treatment effectiveness on categorical scale. Possible responses are:
  0= No screening
  1. Screened for depression with PHQ2 measure
  2. Screened with PHQ2 and meets criteria for further evaluation of depression
  3. Screened and does not meet criteria for further evaluation of depression
Time Frame: End of Treatment (Week 6)
Population: Analysis population consists of all patients providing data at end of treatment.
Measure: Number; unit: participants
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 9 | 2
participants
  No screening | 7 | 2
  Screened by PHQ2 | 2 | 0
  Meets criteria for further evaluation of depressio | 0 | 0
  Does not meet criteria for further evaluation | 0 | 0

31. Other Pre Specified Outcome: Patient's Living Situation at End of Treatment
Description: OASIS question M1100: Patient living situation: This is a measure that combines who lives with the patient and the frequency that assistance is available to them throughout the day. Responses are coded on a 1-15 scale. Measure this as a moderator of treatment effectiveness.
Time Frame: End of Treatment (Week 6)
Population: Analysis population consists of all patients who provided data at end of treatment
Measure: Number; unit: participants
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 9 | 2
participants
  Lives alone | 3 | 0
  Lives with another adult | 3 | 2
  Lives in assisted living | 3 | 0

32. Other Pre Specified Outcome: Caregiver's Ability and Willingness to Assist With ADLs at End of Treatment
Description: OASIS question M2100, item A: Types and sources of assistance for ADLs. Measure as moderator of treatment effectiveness. Responses range from "No assistance needed in this area" to "Assistance needed, but no Caregivers available". Ordinal scale with 6 levels:
  0= No assistance needed
  1. Caregiver provides assistance
  2. Caregiver needs training or support
  3. Caregiver is unlikely to provide assistance
  4. Unclear if caregiver will assist patient
  5. Assistance is needed but is not available
Time Frame: End of Treatment (Week 6)
Population: Analysis population consists of all patients who provided data at end of treatment
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Educational-Medical-Behavioral | Standard Care
Number analyzed (Participants) | 9 | 2
units on a scale | 0 [0 to 1] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 7 month period from baseline visit to 6 month follow-up visit
Description: Adverse events were reported to the study team by the home health care nurses, often as a reason for discontinuation of treatment.
Arm/Group | Educational-Medical-Behavioral | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/8
Other Adverse Events (participants affected / at risk) | 0/11 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Educational-Medical-Behavioral (N=11) | Standard Care (N=8)
Disability (Nervous system disorders) | 0 (0) | 1 (1) — Parkinson's disease, exacerbation

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No